## <u>Title</u>: Pilot Study Testing a Web-Based Moral Elevation Intervention for Veterans with PTSD and Moral Injury <u>ID</u>: D3035-P

NCT: NCT03906240

Principal Investigator: Adam McGuire, Ph.D.

**Statistical Analysis Plan** 

Date: 06.22.2021

## **Statistical Analysis Plan**

All data management and analyses were conducted with R (R Core Team, 2021). To assess the feasibility and acceptability of MOVED, we calculated descriptive statistics for recruitment and retention data, self-report measures that focused on evaluating components of the intervention, and state elevation scores. For all evaluation measures, the mid-point score for a given measure was used as an indicator for adequate feasibility and acceptability (e.g., average/medium levels of acceptability, or higher). The mid-point score for state elevation was also used as an indicator for feasibility to induce elevation.

Qualitative interviews were transcribed, then coded using an inductive approach by two members of the research team and the first author. Two coders reviewed all transcriptions independently, identified codes based on interview responses, then met to discuss and modify codes. A consensus codebook was established and re-applied to all transcriptions. Emergent themes and subthemes were identified by the first author.

Preliminary examination of outcome measures was conducted via paired samples *t*-tests with the base stats package (t.test) and Cohen's *d* effect sizes within each condition with the rstatix package (Kassambara, 2021). Assessment of changes in pre-post measures included all participants who were randomized and provided post-session data.

## References

R Core Team. R: A language and environment for statistical computing. R Foundation for Statistical Computing [Internet]. 2021. Available from: https://www.R-project.org/
Kassambara, A. rstatix: Pipe-Friendly Framework for Basic Statistical Tests [Internet]. 2021.

Available from: https://cran.r-project.org/web/packages/rstatix

Date: 06.22.2021